CLINICAL TRIAL: NCT00504855
Title: Cast Sores With Waterproof Vs. Standard Cast Padding in a Pediatric Population
Brief Title: Cast Sores With Waterproof Vs. Standard Cast Padding
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Staffing changes resulted in the expiration of IRB approval (2/15/12), and recruitment halted (n=84). IRB approval is now current for retrospective analysis.
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Jonathan B. Pellett, Staff Orthopaedic Surgeon, Shriners Hospitals for Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHCH-JPB-1
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Pressure Ulcer
Keywords: Pressure ulcer; Waterproof; Gortex; Cast padding; Pediatric; Heel
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gortex (Waterproof) Cast Padding (Active Comparator): Randomized application of one of two cast padding materials
  Interventions: Other: Casting using Gortex (waterproof) cast padding materials
- Cotton/Cotton-Poly Cast Padding (Active Comparator): Randomized application of one of two cast padding materials
  Interventions: Other: Casting using cotton/cotton-poly cast padding materials

INTERVENTIONS:
Other: Casting using Gortex (waterproof) cast padding materials
  Arms: Gortex (Waterproof) Cast Padding
Other: Casting using cotton/cotton-poly cast padding materials
  Arms: Cotton/Cotton-Poly Cast Padding

SUMMARY:
The purpose of this study is to compare waterproof cast padding material to standard cotton/poly-cotton cast padding material to the presence or absence of cast sores of the heel.

DETAILED DESCRIPTION:
Cast sores result in pain, scarring and sometimes disfigurement. No study has specifically evaluated the efficacy of waterproof cast padding with respect to preventing lower extremity cast sores.

Comparison: Non-blinded randomization to waterproof or cotton/cotton-poly cast padding material in a pediatric population who have lower extremity casts that include the foot and are applied in the operating room. Comparison of cast sore incidence will be made in the two randomized groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient at Shriners Hospital for Children - Honolulu
* Ages 0-18
* Short leg, long leg, spica or Petrie cast that includes the foot
* Cast applied in the operating room

Exclusion Criteria:

* Ponsetti casts (club foot casts with no more surgery than Achilles tenotomy, age < 1 year)
* Splints
* cylinder casts or spicas which don't include the foot

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2007-07; Primary Completion 2012-02 (Actual); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of cast sores, including size, location, grade using Wagner's Classification system for the severe diabetic foot ulcerations | Time of cast application to final cast removal

SECONDARY OUTCOMES:
Presence of: abrasion; pressure/sheer; maceration wetness; infection; cast modification. | Cast application to final cast removal

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan B Pellett, MD, Principal Investigator — Shriners Hospitals for Children, Honolulu; Arabella I Leet, MD, Principal Investigator — Shriners Hospitals for Children, Honolulu
Locations (1):
- Shriners Hospitals for Children - Honolulu, Honolulu, Hawaii, United States

REFERENCES:
- [Background] Wagner FW Jr. Treatment of the diabetic foot. Compr Ther. 1984 Apr;10(4):29-38. No abstract available. PMID 6723248